CLINICAL TRIAL: NCT06188858
Title: Optimal Incision Site Design for Lymphaticovenular Anastomosis in Extremity
Brief Title: Optimal Incision Site Design for Lymphaticovenular Anastomosis in Extremity Lymphedema
Status: Completed | Type: Observational
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Haihua Yang, Chief Physician, Taizhou Hospital
Other Study IDs: Taizhou Hospital OISD
Record Dates: First submitted 2023-12-10; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our aim was to identify optimal incision sites for LVA in extremity lymphedema that would result in the most effective drainage effect for reducing limb edema and enhancing patients' quality of life.

DETAILED DESCRIPTION:
designing the optimal incision sites and identifying functional lymphatic vessels imaging is crucial for success, primarily due to its efficacy in draining edematous lymphatic fluid and reducing swelling in patients with lymphedema. In this study, we conducted patients with LVA lymphedema to investigate the correlation between LVA incision design, intraoperative functional lymphatic vessel assessment, postoperative limb reduction, and patient satisfaction.

question 1：Optimal Incision Site Design for Lymphaticovenular Anastomosis in Extremity lymphedema

ELIGIBILITY:
Inclusion Criteria: Aged 18-80 years; Lymphedema and swelling of the limbs for more than 3 months

-

Exclusion Criteria:

* lipedema；myoedema

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Lymphedema patients
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with lymphedema stage | through study completion, an average of 4 year
  stage 0-3
Number of Optimal Incision Site Design | through study completion, an average of 4 year
  Optimal Incision Site Design for Lymphaticovenular Anastomosis
Rate of lymphatic vessel Functional Parameters | through study completion, an average of 4 year
  intraoperative functional lymphatic vessel assessment
Circumferential Reduction rate | through study completion, an average of 4 year
  postoperative limb reduction and patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: yomao zheng, Study Director — employee; chong liu, Principal Investigator — employee
Locations (1):
- Chong Liu, Zhejiang, China